CLINICAL TRIAL: NCT00216229
Title: A Study Comparing the Effectiveness of Two Different Vaccination Schedules of the Combined Hepatitis A and B Vaccine(Twinrix Adult1440/20)
Brief Title: Twinrix Alternative Schedule Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IDEWE Occupational Health Services (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDEWE-301; 04-033
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2005-12-14 (Estimated); Status verified 2005-09

CONDITIONS: Antibody Response After Vaccination
Keywords: combined hepatitis A and B vaccine; hepatitis B virus; immunity
MeSH Terms: conditions — Hepatitis B | interventions — twinrix

INTERVENTIONS:
Biological: Combined vaccine against hepatitis A and B (Twinrix)

SUMMARY:
To compare the efficiency of protection against hepatitis-B virus by administration of the combined vaccine against hepatitis A and B using the schedule 0-1-12 months against the schedule 0-1-6 months.

1. To compare the seroconversion (>= 1 IU/l) and seroprotection (>= 10 IU/l) rate at month 6,7,12 and 13.
2. To compare the distribution of anti-HBs at these different moments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* a good physical condition as confirmed by history and physical examination at entry of the study;
* for female participants who could become pregnant in the course of the study a contraceptive programme is foreseen;
* all participants have provided written informed consent.

Exclusion Criteria:

* Employees occupationally exposed to hepatitis B virus
* Other exclusion criteria listed for the vaccine (licensed vaccine):
* Each acute disease at the inclusion in the study;
* A history of hypersensibility to one of the components of the vaccine;
* Simultaneous participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-09; Study Completion 2006-02

PRIMARY OUTCOMES:
Anti-HBs antibodies concentration 1 month after 3th vaccine dose

SECONDARY OUTCOMES:
Natural evolution of anti-HBs antibodies concentration between 2nd and 3th vaccine dose (5-11 months)

CONTACTS AND LOCATIONS:
Overall Officials: Antoon A De Schryver, M.D., PhD, Principal Investigator — IDEWE Occupational Health Services
Locations (1):
- IDEWE, Leuven, Belgium